CLINICAL TRIAL: NCT00878358
Title: Hydrotherapy Versus Physiotherapy for Short-term Rehabilitation After Primary TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Leonid Kandel, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hydrotherapy-HMO-CTIL
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Osteoarthritis; Total Knee Replacement
Keywords: Osteoarthritis; Total knee replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Hydrotherapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Active Comparator)
  Interventions: Other: Physiotherapy
- Hydrotherapy (Experimental)
  Interventions: Other: Hydrotherapy

INTERVENTIONS:
Other: Hydrotherapy
  Arms: Hydrotherapy
Other: Physiotherapy
  Arms: Physiotherapy

SUMMARY:
Primary objective:

To compare the effects of short term therapy post total knee replacement (TKR) between a hydrotherapy treatment group and a physiotherapy treatment group.

Secondary objectives:

To compare the effects of short term therapy post total knee replacement (TKR) between a hydrotherapy treatment group and a physiotherapy treatment group based on measurements of timed up and go (TUG, as primary outcome), range of motion, pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for first total knee replacement surgery.

  * Age over 18.
  * Diagnosed with Osteoarthritis.
  * Consent to participate in the trial.

Exclusion Criteria:

* - Rheumatic diseases.
* Neurological diseases involving lower limbs.
* Prior knee surgery in operated knee.
* Secreting surgical wound.
* Skin diseases.
* Incontinence.
* Incapable of signing informed consent.
* Patients living outside Jerusalem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 6 weeks

SECONDARY OUTCOMES:
Oxford knee score | 6 weeks
Visual analogue pain score | 6 weeks
Range of knee motion | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel